CLINICAL TRIAL: NCT05540574
Title: Randomized Placebo-Controlled Crossover Trial of Zolpidem for Sleep in Children With Autism
Brief Title: Trial of Zolpidem for Sleep in Children With Autism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB-67221; 1P50HD109861 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: zolpidem; sleep; clinical trial; autism
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zolpidem, then Placebo (Experimental): Participants will first receive Zolpidem for a 4-week period. A 5 mg dose of Zolpidem will be given at bedtime for one week and then will increase to 10 mg if needed and if well tolerated.
  Participants will then receive Placebo (fake tablet) for a 4-week period. A 5 mg dose of matching Placebo will be given at bedtime for one week and then will increase to 10 mg if needed and if well tolerated.
  Interventions: Drug: Zolpidem; Drug: Placebo
- Placebo, then Zolpidem (Experimental): Participants will first receive Placebo (fake tablet) for a 4-week period. A 5 mg dose of matching Placebo will be given at bedtime for one week and then will increase to 10 mg if needed and if well tolerated.
  Participants will then receive Zolpidem for a 4-week period. A 5 mg dose of Zolpidem will be given at bedtime for one week and then will increase to 10 mg if needed and if well tolerated.
  Interventions: Drug: Zolpidem; Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem — 5mg (and up to10mg) Diphenhydramine given orally
  Other Names: Ambien
Drug: Placebo — Matching Placebo given orally

SUMMARY:
The purpose of this study is to examine the effect of zolpidem on sleep in children and adolescents with Autism Spectrum Disorder (ASD). Zolpidem is a nonbenzodiazepine GABAa receptor agonist drug that acts as a hypnotic. To accomplish this, the investigators will use a randomized double-blind placebo-controlled crossover 8-week study design to examine the effect of zolpidem on sleep physiology as assessed by polysomnography (PSG), actigraphy, circadian rhythm, and clinical measures.

ELIGIBILITY:
Inclusion criteria:

Participants will meet the following

* Outpatients between 8 and 17 years of age with only 12- 17 years of age at time of consent during year 1
* Diagnostic and Statistical Manual, 5th edition (DSM-5) criteria for Autism Spectrum Disorder (ASD) on the basis of clinical evaluation, confirmed with the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule, 2nd Ed (ADOS-2)
* Males and females
* Availability of polysomnography (PSG) and/or actigraphy data
* Sleep disturbances as assessed using Children's Sleep Habits Questionnaire (CSHQ) with a score of 41 or higher and sleep efficiency of 85% or less and/or total sleep time less than 7 hours and/or wake after sleep onset of more than 30 minutes as measured by polysomnography (PSG) or actigraphy.
* care provider who can reliably bring participant to clinic visits, provide trustworthy ratings, and interacts with participant on a regular basis
* stable medications for at least 2 weeks, with the exception of Prozac which is required to be stable for at least 4 weeks
* no planned changes in psychosocial and biomedical interventions during the trial
* willingness to provide additional saliva samples and participate in key study procedures (i.e., safety measurements every visit, PSG at weeks 4 and 8, and wear the actigraphy watch for 2 weeks before the beginning of trial as well as during the 8 weeks of the trial)
* requirement of dual protection contraception use in females who are sexually active and are of childbearing potential. Dual use contraceptive methods involve the use of both a hormonal method (oral contraceptives, long-acting reversible contraceptives, etc.) and a barrier method (condoms).

Exclusion criteria:

Participants will be excluded if one or more of the following is met

* active suicidal ideation or DSM-5 diagnosis of severe depression, substance use disorder, schizophrenia, schizoaffective disorder, or psychotic disorder
* unstable medical problems: migraine, asthma, seizure disorder, significant physical illness (e.g., anaphylaxis, serious liver, renal, or cardiac pathology) and hepatic insufficiency
* evidence of a metabolic, or infectious etiology for the participant's autism on the basis of medical history, neurologic history, and available tests for inborn errors of metabolism;
* pregnant or sexually active females not using a reliable method of contraception (urinary tests for pregnancy will be employed in this study)
* individuals taking beta-blockers (local or systemic), benzodiazepines, antiepileptic medications, melatonin, antihistamines and antidepressants
* history of hypersensitivity to zolpidem
* history of severe side effects from zolpidem
* history of adequate trial of zolpidem
* current use of any medications known to interact with zolpidem such as medications inhibiting CYP3A4 and CYP1A2
* history of complex sleep-related behaviors
* individuals using alcohol, marijuana and other substances.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in sleep architecture as measured by polysomnography (PSG), examples include sleep latency and non-rapid eye movement (NREM) | Baseline, Week 4 and Week 8

SECONDARY OUTCOMES:
Change from baseline in sleep efficiency as measured by actigraphy | Baseline, Week 4 and Week 8

OTHER OUTCOMES:
Change from baseline on Children's Sleep Habits Questionnaire (CSHQ) subscale score | Baseline, Week 4 and Week 8
Change from baseline on Aberrant Behavior Checklist, Second Edition (ABC-2) subscale scores | Baseline, Week 4 and Week 8
Change from baseline on Parent Sleep Habits Questionnaire Parent (PSHQ) scores | Baseline, Week 4 and Week 8
Change from baseline on Clinical Global Impression Scale (CGI) scores | Baseline, Week 4 and Week 8
Change from baseline on Child Behavior Checklist (CBCL) scores | Baseline, Week 4 and Week 8
Change from baseline on Social Responsiveness Scale, Second Edition (SRS-2) scores | Baseline, Week 4 and Week 8
Change from baseline on Repetitive Behavior Scale - Revised (RBS-R) scores | Baseline, Week 4 and Week 8
Change from baseline on Sensory Profile Questionnaire (SPQ) scores | Baseline, Week 4 and Week 8
Change from baseline on Stanford Social Dimension Scale (SSDS) scores | Baseline, Week 4 and Week 8
Change from baseline on Dimensional Assessment of Repetitive Behaviors (DARB) scores | Baseline, Week 4 and Week 8
Change from baseline on NEuroPSYchological Assessment, 2nd Edition (NEPSY-2) Affect Recognition scores | Baseline, Week 4 and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit de-identified clinical data to the NIMH Data Archive (NDA) data repository.
URL: https://nda.nih.gov/nda/data-contribution.html